CLINICAL TRIAL: NCT05650450
Title: A Hybrid Approach Evaluating A Drug-Coated Balloon in Combination With A New Generation Drug-Eluting Stent in the Treatment of Long Diffuse Coronary Artery Disease: The HYPER II Study
Brief Title: Drug-Coated Balloon in Combination With New Generation Drug-Eluting Stent in the Treatment of Long Diffuse Coronary Artery Disease
Acronym: HYPER II
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: HYPER II
Record Dates: First submitted 2022-12-04; First posted 2022-12-14 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with diffuse CAD disease treated with hybrid strategy (DES+DCB)
  Interventions: Device: DES+DCB

INTERVENTIONS:
Device: DES+DCB — Hybrid approach is defined as overlapping or slightly (2-3 mm) superimposing a new generation DES for a de novo long (>38 mm) lesion (located in the larger, more proximal part of the vessel -reference vessel diameter -RVD >2.75 mm-) and DCB inflation for a concomitant and contiguous de novo small vessel disease (distally located with RVD ≤2.75 mm ≥ 2.0 mm)

SUMMARY:
An observational study to evaluate safety and efficacy of the hybrid approach DES/DCB in the treatment of long diffuse de novo coronary artery disease

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm, multi-center study aiming to assess the feasibility and the clinical outcomes of using the Restore DCB (Cardionovum GmbH, Bonn, Germany) in combination ("hybrid approach") with a new generation DES (type at operator's discretion) for the treatment of diffuse CAD (Coronary Artery Disease) encountered in daily clinical practice (lesion length > 38 mm). The rationale of the proposed strategy derives from the characteristics of DCB in treating the atherosclerotic disease without leaving a permanent structure in the vessel especially in case of diffuse CAD -avoiding a long metallic, permanent cage within extended coronary segments

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with stable or unstable CAD eligible for PCI (according to the international guidelines) because of diffuse long (>38 mm) CAD involving contiguous segments of the same vessel suitable for a hybrid approach (RVD>2.75 mm in the proximal DES target segment and RVD ≤2.75 mm ≥ 2.0 mm for the distal DCB target segment);
* Signed Patient Informed Consent/Data Release Form

Exclusion Criteria:

* Age <18 years;
* Cardiogenic shock;
* Pregnancy or breastfeeding;
* Target vessel reference diameter (within planned device deployment segments) <2.0 or >5.0 mm;
* Comorbidities with life expectancy <12 months
* Severe calcification or/tortuosity proximally or at the DCB target segment;
* Prior PCI and stent implantation in the target vessel.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting with stable or unstable CAD eligible for PCI (according to the international guidelines) because of diffuse long (>38 mm) CAD involving contiguous segments of the same vessel suitable for a hybrid approach (RVD>2.75 mm in the proximal DES target segment and RVD ≤2.75 mm ≥ 2.0 mm for the distal DCB target segment). Hybrid approach is defined as overlapping or slightly (2-3 mm) superimposing a new generation DES in the larger, more proximal part of the vessel -reference vessel diameter -RVD >2.75 mm- and DCB inflation for a concomitant and contiguous de novo small vessel disease - distally located with RVD ≤2.75 mm ≥2.0 mm.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
TLF in DES/DCB treated segment at 12 months | 12 months
  Target lesion failure (TLF) defined as a composite of cardiac death, target vessel myocardial infarction (TV-MI) and ischemia-driven target lesion revascularization (ID-TLR) in the DES- and/or the drug-coated balloon (DCB)-treated segment within 12 months after the index procedure

SECONDARY OUTCOMES:
Procedural success | At procedure
  Procedural success defined as both DCB/DES delivery and implantation at the "target" lesion site with <30% diameter stenosis (DS) in the DCB-treated segment and <10% DS in the DES-treated segment and distal TIMI (Thrombolysis in Myocardial Infarction) 3 flow
Peri-procedural myocardial infarction | Pre-discharge
  Peri-procedural myocardial infarction defined as an elevation of cardiac biomarkers (troponin or creatine kinase-myocardial band) >3 times the upper limit of normal
TLF | Pre-discharge, 30 days, 12 months, 24 months
  TLF and its singular components (cardiac death, any TV-MI excluding peri-procedural MI, ID-TLR)
Thrombosis | In-hospital (within 7 days after PCI), at 30-days, 12 months, 24 months follow-up
  Any definite/probable DES- or DCB-treated segment thrombosis
Flow-limiting dissection | At procedure
  low-limiting dissection (type C-F waiting 3 minutes after DCB inflation) requiring additional DES implantation in the DCB-treated segment

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico S.Ambrogio, Milan, Italy

REFERENCES:
- [Background] Ielasi A, Buono A, Pellicano M, Tedeschi D, Loffi M, Donahue M, Regazzoli D, De Angelis G, Danzi G, Reimers B, Tespili M. A HYbrid APproach Evaluating a DRug-Coated Balloon in Combination With a New-Generation Drug-Eluting Stent in the Treatment of De Novo Diffuse Coronary Artery Disease: The HYPER Pilot Study. Cardiovasc Revasc Med. 2021 Jul;28:14-19. doi: 10.1016/j.carrev.2020.07.036. Epub 2020 Jul 31. PMID 32933874
- [Background] Ielasi A, Miyazaki T, Geraci S, Testa L, Abdel-Wahab M, Kawamoto H, Ruparelia N, Sato T, Caramanno G, Bedogni F, Tespili M, Colombo A, Latib A. Hybrid strategy with a bioresorbable scaffold and a drug-coated balloon for diffuse coronary artery disease: the "no more metallic cages" multicentre pilot experience. EuroIntervention. 2016 Apr 8;11(14):e1589-95. doi: 10.4244/EIJV11I14A309. PMID 27056119